CLINICAL TRIAL: NCT00522470
Title: Effects of Rosiglitazone on Serum Ghrelin and Peptide YY Levels in Diabetic Women
Brief Title: Effects of Rosiglitazone on Serum Ghrelin and Peptide YY Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KA 06/299
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
We aimed to evaluate the effects of rosiglitazone on serum ghrelin and peptide yy levels in diabetic women.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed, drug naive women with type 2 diabetes

Exclusion Criteria:

* presence of severe cardiovascular disease (eg, New York Heart Association class III or IV congestive heart failure or a history of myocardial infarction or stroke)
* presence of thyroid, pituitary, nutritional, hepatic, renal, or neoplastic disorders

Ages: 45 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Berberoglu, MD, Principal Investigator — Baskent University Faculty of Medicine
Locations (1):
- Baskent University Hospital Department of Endocrinology, Ankara, Bahçelievler, Turkey (Türkiye)

REFERENCES:
- [Derived] Berberoglu Z, Yazici AC, Bayraktar N, Demirag NG. Rosiglitazone decreases fasting plasma peptide YY3-36 in type 2 diabetic women: a possible role in weight gain? Acta Diabetol. 2012 Dec;49 Suppl 1:S115-22. doi: 10.1007/s00592-011-0352-3. Epub 2011 Nov 19. PMID 22101910